CLINICAL TRIAL: NCT04605237
Title: Detection, Treatment and Survival of Pancreatic Cancer Recurrence in the Netherlands
Brief Title: Pancreatic Cancer Recurrence in the Netherlands
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: Amsterdam UMC, location VUmc (Other); Erasmus Medical Center (Other); Catharina Ziekenhuis Eindhoven (Other); Radboud University Medical Center (Other); University Medical Center Groningen (Other); Jeroen Bosch Ziekenhuis (Other); Leiden University Medical Center (Other); Maastricht University Medical Center (Other); Maasstad Hospital (Other); Amphia Hospital (Other); Onze Lieve Vrouwe Gasthuis (Other); Reinier de Graaf Groep (Other); Isala (Other); St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Prof. dr. I.Q. Molenaar, MD, PhD, Prof. dr., UMC Utrecht
Other Study IDs: 18-036/C
Record Dates: First submitted 2020-10-15; First posted 2020-10-27 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Pancreatic Cancer; Pancreas Cancer; PDAC
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this nationwide, observational cohort study is to evaluate current surveillance strategies after primary resection of pancreatic ductal adenocarcinoma (PDAC) in the Netherlands, with regard to the detection, treatment and survival of PDAC recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a pancreatic resection (PPPD, Whipple, distal pancreatectomy or total pancreatectomy) for histologically proven PDAC in one of the 16 Dutch centers for pancreatic surgery

Exclusion Criteria:

* Patients with 30-day postoperative mortality

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients registered within the prospective, mandatory Dutch Pancreatic Cancer Audit who underwent resection of histologically proven PDAC.
Sampling Method: Non-Probability Sample
Enrollment: 1750 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of PDAC recurrence | Within a follow-up period up to 5 years
  Incidence of PDAC recurrence within the Netherlands; PDAC recurrence is either pathologically proven, or suspected through cross-sectional imaging, preferably confirmed by consensus during a multidisciplinary meeting.
Patterns of PDAC recurrence | Within a follow-up period up to 5 years
  * Asymptomatic vs. symptomatic: Symptomatic recurrence is defined as the presence of symptoms suggestive for PDAC recurrence at recurrence diagnosis. If PDAC recurrence is detected in absence of suspected symptoms, disease recurrence was defined as asymptomatic.
  * First site of recurrence: isolated local recurrence, liver-only, lung-only, multiple-site, other isolated distant
  * Early vs. late recurrence: disease-free survival ≥12 months vs. <12 months
Treatment of PDAC recurrence | Within a follow-up period up to 5 years
  Either systemic and/or local treatment or best-supportive-care
Survival | Within a follow-up period up to 5 years
  Overall survival (from the time of resection), disease-free survival (from the time of resection), post-recurrence survival (from the time of recurrence diagnosis)

SECONDARY OUTCOMES:
Presence of symptoms at time of (suspected) recurrence | Within a follow-up period up to 5 years
  Which symptoms are associated with PDAC recurrence?
Performance score at time of recurrence detection | Within a follow-up period up to 5 years
  What is the ECOG performance score of patients at time of recurrence diagnosis?
Use of imaging procedures during follow-up | Within a follow-up period up to 5 years
  How much imaging procedures are performed during postoperative follow-up for the detection of PDAC recurrence? Are these procedures routinely performed?
Number of histologically confirmed recurrences | Within a follow-up period up to 5 years
  How often is PDAC recurrence histologically confirmed?

CONTACTS AND LOCATIONS:
Overall Officials: I. Quintus Molenaar, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-29): https://cdn.clinicaltrials.gov/large-docs/37/NCT04605237/Prot_SAP_000.pdf